CLINICAL TRIAL: NCT05802797
Title: Bioavailability and Pharmacodynamics of Eicosapentaenoic Acid and Docosahexaenoic Acid in Soymilk and Commercial Supplements
Brief Title: Bioavailability and Pharmacodynamics of EPA and DHA From Fortified Soymilk and Capsules
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Yael Vodovotz, Professor, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: OSU-87
Record Dates: First submitted 2023-03-22; First posted 2023-04-07 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Healthy Diet
Keywords: Algae Oil; EPA and DHA; Omega-3 Fatty Acids

STUDY DESIGN:
Intervention Model Description: 24 participants (12 men and 12 women) will be randomized to two intervention groups.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algae Oil Fortified Soymilk (Experimental): Subjects will drink 12 ounces of 0.4% algae oil-fortified soymilk
  Interventions: Other: Algae Oil Fortified Soymilk
- Algae Oil Supplements (Active Comparator): Subjects will take 2 commercial algae oil capsules.
  Interventions: Dietary Supplement: Algae Oil Capsule

INTERVENTIONS:
Other: Algae Oil Fortified Soymilk — Flavored soymilk beverage fortified with 0.4% algae oil with both EPA and DHA
  Arms: Algae Oil Fortified Soymilk
Dietary Supplement: Algae Oil Capsule — Algae oil capsules with EPA and DHA
  Arms: Algae Oil Supplements

SUMMARY:
This study will compare the algae oil fortified soymilk to a commercial algae oil capsule containing the same base oil with the goal of demonstrating equivalent or greater accumulation of EPA and DHA in blood lipid pools.

DETAILED DESCRIPTION:
Research shows that fish oil and its component fatty acids EPA and DHA provide health benefits such as reducing the risk of cardiac death and lowering inflammation. Yet a large portion of the population is not consuming the recommended amount of fish due to high cost, dietary restrictions such as vegetarianism/veganism, concerns about high levels of mercury, general dislike, and other factors. Additionally, to meet the recommendations fish and fish oil production present sustainability challenges. A potential alternative is to utilize EPA and DHA from algae. These sustainable oils can be added to foods increasing the potential for fatty acids to counteract chronic disease and increasing access to general consumers. Previously, our lab has developed, and optimized EPA and DHA fortified non-dairy plant milk beverages utilizing algae oil emulsions (food grade). Up to 0.4% algae oil can be added to soymilk with limited changes to overall liking. This study will compare the algae oil fortified soymilk to a commercial algae oil capsule containing the same base oil with the goal of demonstrating equivalent or greater accumulation of EPA and DHA in blood lipid pools. Subjects will consume either one beverage or two capsules per day, containing equivalent amounts of EPA and DHA. Blood will be taken at 4 time points throughout the 6 week study, every two weeks and analyzed for EPA and DHA in different lipid types. Additionally, participants will complete a food frequency questionnaire to evaluate their normal diet, sensory evaluation (overall liking, and attribute evaluation) of the beverages, and daily symptom and intake logs to track consumption and any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 30 kg/m2

Exclusion Criteria:

* Being pregnant or nursing
* Having anemia or a condition that influences the ability to donate blood safely
* Allergies to the beverage or pill ingredients
* Diabetes
* High triglycerides or cholesterol
* Coagulation disorder
* Anticoagulation therapy or any drug that affects blood clotting.
* Taking prescribed dietary omega-3 fatty acid medications including fish oil or algae oil within the last 3 months
* Taking non-prescribed dietary omega-3 fatty acid supplements within the last 3 months and not willing to discontinue taking them for the study period
* Taking lipid lowering medications such as statins
* Sensory impairments which affect ability to taste, smell, or see food products

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Erythrocyte EPA and DHA levels | 4 weeks
  Percent EPA and DHA of total fatty acids in erythrocyte samples

SECONDARY OUTCOMES:
Plasma EPA and DHA levels | 4 weeks
  Percent EPA and DHA of total fatty acids in plasma samples
Peripheral blood mononuclear cell (PBMC) EPA and DHA levels | 4 weeks
  Percent EPA and DHA of total fatty acids in PBMC samples

OTHER OUTCOMES:
Compliance | 4 weeks
  Percent of days that participants consume their beverage or pill

CONTACTS AND LOCATIONS:
Overall Officials: Yael Vodovotz, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05802797/Prot_000.pdf
  • Informed Consent Form (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT05802797/ICF_001.pdf